CLINICAL TRIAL: NCT05045586
Title: Modified Coronally Advanced Tunnel With Cross-linked Hyaluronic Acid in Addition to Connective Tissue Graft Compared With Subepithelial Connective Tissue Graft Alone for Treatment of Multiple Gingival Recession: Randomized Clinical Trial
Brief Title: MCAT With HA and sCTG Compared With sCTG Alone for Treatment of Multiple Gingival Recession: Clinical Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WUM.Perio.03
Record Dates: First submitted 2021-09-06; First posted 2021-09-16 (Actual); Last update posted 2021-10-12 (Actual); Status verified 2021-06

CONDITIONS: Gingival Recession
Keywords: connective tissue graft; tunneling flap procedure; hyaluronic acid
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Modified Coronally Advanced Tunnel With Connective Tissue Graft (Experimental): Procedure: A modified microsurgical tunnel technique by Zuhr et al. (2007). Initial sulcular incisions with a microsurgical blade are followed by a split-thickness buccal flap preparations using the tunneling knives. The preparation is extended into the mucosal tissue to gain sufficient flap mobility. The papillary regions are detached in their buccal aspects with the periosteum. The graft is inserted into the tunnel and stabilized with absorbable suspensory sutures. The buccal flap is advanced coronally and stabilized with non-absorbable suspensory sutures.
  Interventions: Device: The tunnel technique for root coverage with CTG without Cross-linked Hyaluronic Acid
- MCAT With Cross-linked Hyaluronic Acid in Addition to CTG (Active Comparator): Procedure: A modified microsurgical tunnel technique by Zuhr et al. (2007). Initial sulcular incisions with a microsurgical blade are followed by a split-thickness buccal flap preparations using the tunneling knives. The preparation is extended into the mucosal tissue to gain sufficient flap mobility. The papillary regions are detached in their buccal aspects with the periosteum. The root surfaces are applied with cross-linked hyaluronic acid. The graft is inserted into the tunnel and stabilized with absorbable suspensory sutures. The buccal flap is advanced coronally and stabilized with non-absorbable suspensory sutures.
  Interventions: Device: The tunnel technique for root coverage with CTG andCross-linked Hyaluronic Acid

INTERVENTIONS:
Device: The tunnel technique for root coverage with CTG without Cross-linked Hyaluronic Acid — The tunnel technique for root coverage with CTG without Cross-linked Hyaluronic Acid
  Arms: Modified Coronally Advanced Tunnel With Connective Tissue Graft
Device: The tunnel technique for root coverage with CTG andCross-linked Hyaluronic Acid — The tunnel technique for root coverage with CTG andCross-linked Hyaluronic Acid
  Arms: MCAT With Cross-linked Hyaluronic Acid in Addition to CTG

SUMMARY:
Microsurgical tunneling flap procedures using connective tissue grafts (CTG) are predictable for treating teeth with gingival recessions. Cross-linked hyaluronic acid can be used in conjunction with subepithelial palatal connective tissue grafts to improve postsurgical results. The aim of this study is to evaluate clinically the use of tunnel technique with CTG and cross-linked hyaluronic acid in addition to CTG alone for the treatment of multiple gingival recessions.

DETAILED DESCRIPTION:
The treatment of multiple adjacent recession appears to be challenging for the clinician due to large surgical field, variation in teeth position in the dental arch (prominent roots), variation in recession size, thin phenotype and insufficient keratinized tissue in many teeth. Surgical treatment of all multiple recession in one dental arch during one session appears to be optimum. Surgical treatment time is longer, however patient doesn't need to undergo multiple surgeries, pharmacological therapies and postsurgical instructions. Esthetic concern seems to be one of the most common complaints from patients. Among utilized surgical techniques tunneling flap procedures using connective tissue grafts (CTG) with or without biologics such as an enamel matrix derivative (EMD) or hyaluronic acid (HA) provided the most successful outcomes for the treatment. Cross-linked hyaluronic acid can be used in conjunction with subepithelial palatal connective tissue grafts to improve postsurgical results and improving healing process. The aim of this study is to evaluate clinically the use of tunnel technique with CTG and cross-linked hyaluronic acid in addition to CTG alone for the treatment of multiple gingival recessions.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Bilateral multiple gingival recessions in homologous teeth

Exclusion Criteria:

* Full-mouth plaque index ≥ 20% (Ainamo & Bay 1975)
* Full-mouth sulcus bleeding index ≥ 15% (Mühlemann & Son 1971)
* Smoking
* Systemic diseases with compromised healing potential of infectious diseases
* Drugs affecting periodontal health / healing
* Pregnant and lactating females
* Previous periodontal surgery in the area

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2021-09-15 (Actual); Primary Completion 2022-09-15 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Periodontal parameters measured before surgery. | 1-7 days before surgery
  1. Probing pocket depth (PPD) MEASURED IN MILIMETERS: distance from the gingival margin to the bottom of the gingival sulcus
  2. Clinical attachment level (CAL) MEASURED IN MILIMETERS: distance from the cementoenamel junction to the bottom of the gingival sulcus
  3. Recession height (RH) MEASURED IN MILIMETERS: distance from the cementoenamel junction to the gingival margin
  4. Width of keratinized tissue (WKT) MEASURED IN MILIMETERS: distance between the most apical point of the gingival margin and the mucogingival junction
  5. Gingival thickness (GT) MEASURED IN MILIMETERS: thickness of the gingiva measured 2-3 mm apical to the gingival margin

SECONDARY OUTCOMES:
Periodontal parameters measured after surgery. | 12 months after surgery
  1. Probing pocket depth (PPD): distance from the gingival margin to the bottom of the gingival sulcus
  2. Clinical attachment level (CAL): distance from the cementoenamel junction to the bottom of the gingival sulcus
  3. Recession height (RH): distance from the cementoenamel junction to the gingival margin
  4. Width of keratinized tissue (WKT): distance between the most apical point of the gingival margin and the mucogingival junction
  5. Gingival thickness (GT): thickness of the gingiva measured 2-3 mm apical to the gingival margin
  ALL ABOVE PARAMETERS ARE MEASURED IN MILIMETERS

OTHER OUTCOMES:
Patient-reported outcomes based on VAS scales | 2 weeks after surgery
  Questionnaires:
  Scale 1: Pain after surgery (during recent 2 weeks) from 0 (no pain) to 10 (very big pain)

CONTACTS AND LOCATIONS:
Overall Officials: Batlomiej Górski, PhD, Principal Investigator — Department of Periodontology and Oral Mucosa Diseases, Medical University of Warsaw
Locations (1):
- Department of Periodontology and Oral Mucosa Diseases, Medical University of Warsaw, Warsaw, Mazowsze, Poland

REFERENCES:
- [Derived] Gorski B, Skierska IM, Gelemanovic A, Roguljic M, Bozic D. Multiple Recessions Coverage Using the Modified Tunnel Technique and Connective Tissue Graft with or Without Cross-Linked Hyaluronic Acid: 2-Year Outcomes of RCT. J Funct Biomater. 2025 Mar 4;16(3):87. doi: 10.3390/jfb16030087. PMID 40137366
- [Derived] Gorski B, Skierska IM, Nijakowski K, Brodzikowska A. Tunnel Technique and Subepithelial Connective Tissue Graft, With or Without Cross-Linked Hyaluronic Acid, in the Treatment of Multiple Gingival Recessions: Prognostic Parameters for Clinical Treatment Outcomes of Randomized Controlled Trial. J Clin Med. 2024 Nov 10;13(22):6758. doi: 10.3390/jcm13226758. PMID 39597902